CLINICAL TRIAL: NCT06968884
Title: Enhanced Recovery After Surgery for Patients With Sarcoma of the Extremities and Trunk.
Brief Title: Application of a Comprehensive Protocol Aimed at Reducing the Risk of Complications After Surgery for Sarcoma. Interventions Before, During and After Surgery for Known and Presumed Risk Factors Compared to Standard of Care in a Total of 300 Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00847-01; K2024-9009 (Other: Karolinska university Hospital); RA 2024/98 (Other: Karolinska Institutet)
Record Dates: First submitted 2025-04-14; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Surgical Complications; Sarcoma
Keywords: risk reduction; eras
MeSH Terms: conditions — Sarcoma; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Interventional prospective study. Control group included first and interventional group included thereafter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group - best available care (Active Comparator): Patients receive best available care. Sarcoma surgery, transfusions and medication given is best known to medical professionals in care.
  Interventions: Procedure: Control (Standard treatment)
- ERAS intervention (Active Comparator): The complete protocol including pre- per- and postop adjustments in addition to sarcoma surgery.
  Interventions: Other: Protocol based

INTERVENTIONS:
Other: Protocol based — Preoperative administration of iron, b12 and folate if criteria is met. Medication to aid in smoking cessation is offered if patient uses tobacco. Nutritional supplements offered pre-operative is patient malnurished and preoperative drink offered to all.
  Anaesthetic method adapted with increased use of epidural, blocks and local anaesthesia.
  Administration on TXA and fluids according to protocol. Postoperative nutritional drink to increase protein intake. Early mobilisation to reduce risk of VTE.
  Arms: ERAS intervention
Procedure: Control (Standard treatment) — Preoperative bloods including haemoglobin to establish that surgery is safe. Transfusions given if clinically necessary, no other protocol for anaemia treatment other then available clinical guidelines.
  Peri- and postoperative treatment given in accordance with best clinical practice, no additional protocol.
  Arms: Control group - best available care

SUMMARY:
Sarcoma is a rare malignancy made up by several sub types that can occur throughout the body. Roughly speaking, the division into soft tissue sarcoma (STS) and skeletal sarcoma (SS) can be made. STS of the limbs and trunk are primarily treated by surgical removal of the tumour and a margin of surrounding healthy tissue. Since size, depth and locale of tumours vary widely, surgery is seldom standardised.

Both STS and SS commonly result in large resections, leaving tissue defects that are prone to local complications such as seroma formation, wound dehiscence and infection. A wound complication following surgery can be considered minor if it does not call for additional surgery, i.e. seroma formation, a superficial infection or delayed wound closure that can be helped by oral antibiotics or wound care. A major wound complication is one that requires surgical treatment like debridement surgery, secondary suture of a ruptured wound or flap-reconstruction.

It is known that some tumour related factors increase the risk of wound complications, e.g. certain anatomical areas such as the inner thigh, large size and higher grade of the tumour. Other patient related factors known to influence the risk of complication are smoking, malnutrition and diabetes.

There is some research on orthopaedic patients looking at intraoperative factors that could affect risk of infection. Time in surgery, prophylactic antibiotics and bleeding have all been shown to influence outcome.

Enhanced Recovery After Surgery (ERAS) is a project implemented in other fields of surgery. It is a complete take on the risk factors for complications surrounding a patient and their surgery, as well as recovery afterwards. Some patient-related (intrinsic) risk factors associated with complications, such as obesity and alcohol abuse, take time to change. In other cases, even a short duration of for example smoke-cessation, correction of anaemia or better nutrition could have an effect on results. Intraoperative environmental (extrinsic) adjustments like surgical haemostasis and administration of Tranexamic acid are known to reduce risk of haematoma formation. This in turn reduces both the need for transfusion and the risk of infection.

In other areas, multimodal anaesthesia and analgesia have been shown to decrease use of opioids while still offering sufficient pain relief. This leads to reduced postoperative nausea and further promotes early postoperative mobilisation.

The thought behind a structured program addressing risk factors before, during and after surgery being that the collective risk reduction will big enough to be measurable where individual efforts might not be.

Since sarcoma surgery is burdened by postoperative complications, every possibility to affect this should be explored.

DETAILED DESCRIPTION:
Prospective inclusion of patients 15 years or older, undergoing surgery for STS or SS. These include grade 1-3 sarcomas and all types of resection and reconstruction. The first 150 patients are the control group, treated according to standard procedure (best available care). The following 150 patients are the ERAS-interventions group.

This protocol with consecutive and not parallel arms is designed because of the difficulty to implement a new standard of care. To do so in only part of the population would increase the risk of contamination between groups and make evaluation harder.

Preoperative labs for anaemia and nutritional status are drawn at suspicion of sarcoma at the first visit to clinic. Patient reported information on smoking, alcohol use, weight and physical activity are registered. Preoperative interventions such as the administration of parenteral iron, enteral B1 or Folic acid, medication for smoking cessation or nutritional complements are prescribed.

The extra costs for nutritional supplements, iron injection and blood tests are minor. If number of days in hospital is shortened or any complication avoided these costs will be negligible.

Hypotheses A structured pre-, per- and postoperative effort on minimising known risk factors for complications are believed to reduce the rate of such complications by 40% compared to patients treated traditionally.

Primary outcome

* Early (<30 days) postoperative complications. Secondary outcomes
* Delayed complications (30d-1y), time to wound healing, time in hospital, death and patient reported outcome measures using EQ5d.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoma of the extremities or trunk
* Surgery for sarcoma at karolinska university Hospital in Sweden
* Age 15 years or older

Exclusion Criteria:

* Not meeting inclusion
* Patient declines
* Patient not a Swedish citizen

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication | 30 days postoperative
  Defined as venous trombo-embolism (VTE) or a local wound complication at 30 days postoperative. Complication severity sub typed using the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Delayed complications (30d-1y) | 30 days to 1 year postoperative
  Complications that are not in the immediate postoperative period, byt appear 1-12 months after surgery. This will include surgical wound complications resulting in need for additional surgery, time in hospital and death. Clavien-Dindo classification is used to stratify severity.

OTHER OUTCOMES:
Patient reported outcome measures (PROMS) | 1 year postoperative
  The form EQ5D (EuroQol 5 dimensions) is filled out by patients at 1 year postoperative. Questions regarding patients' level of mobility, self-care, usual activities, pain and discomfort, and anxiety and depression are answered. Each generates a number 1-5 where 1 indicates no problem and 5 is most severe.
  The possible outcomes vary from 5-25 (11111 and 55555) where a higher number indicates worse self reported health.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Tsagkozis, Associate professor, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Summarised data, text, tables and figures can be shares. Protocols and interventions as well. This data is available for up to 5 years after publication.

REFERENCES:
- [Background] White JJ, Houghton-Clemmey R, Marval P. Enhanced recovery after surgery (ERAS): an orthopaedic perspective. J Perioper Pract. 2013 Oct;23(10):228-32. doi: 10.1177/175045891302301004. PMID 24279038
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Perrault DP, Lee GK, Yu RP, Carre AL, Chattha A, Johnson MB, Gardner DJ, Carey JN, Tseng WW, Menendez LR, Wong AK. Risk Factors for Wound Complications After Soft Tissue Sarcoma Resection. Ann Plast Surg. 2021 Mar 1;86(3S Suppl 2):S336-S341. doi: 10.1097/SAP.0000000000002592. PMID 33234885
- [Background] Moore J, Isler M, Barry J, Mottard S. Major wound complication risk factors following soft tissue sarcoma resection. Eur J Surg Oncol. 2014 Dec;40(12):1671-6. doi: 10.1016/j.ejso.2014.10.045. Epub 2014 Oct 18. PMID 25456440